CLINICAL TRIAL: NCT05450055
Title: A Randomized Controlled Trial to Investigate Effect of Postoperative Intraperitoneal Lidocaine on the Analgesic and Prognosis of Patients With Ovarian Cancer
Brief Title: Intraperitoneal Lidocaine in Ovarian Cancer Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M2021589
Record Dates: First submitted 2022-05-31; First posted 2022-07-08 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Ovarian Cancer; Post Operative Pain
Keywords: Postoperative intraperitoneal lidocaine; Intraperitoneal analgesic; Ovarian cancer; Prognosis
MeSH Terms: conditions — Ovarian Neoplasms; Pain, Postoperative | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Sixty patients were expected to participate in a centralized randomized study method divided into two groups of 30 patients per group: the intraperitoneal analgesic group and the normal saline control group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intraperitoneal analgesic group (Experimental): Before the end of surgery, patients in the experimental group (L group) were extensively sprayed with 20mL (100mg) 0.5% lidocaine intraperitoneally before the peritoneum was sutured. The surgeon placed intraperitoneal catheter with the catheter tip above the vaginal end while placing percutaneous drainage tube. Patients in both groups were routinely given flurbiprofen axel 50mg intravenously for analgesia. Local infiltration anesthesia was performed with 20mL 1% lidocaine at the incision area. The intraperitoneal catheter was connected to the electronic analgesia pump, and the infusion of 0.5% lidocaine 10mL/h was interrupted from 1 to 72h after surgery, with a total volume of 720mL in the pump. At the same time, patients in both groups were connected with intravenous controlled intravenous controlled analgesia (PCIA) : sufentanil 100µg to 100mL normal saline, background dose of 2mL/h, single push injection of 0.5mL, locked for 15 minutes.
  Interventions: Procedure: intraperitoneal lidocaine analgesic or normal saline as control
- control group (Placebo Comparator): Before the end of surgery, patients in the control group (C group) were extensively sprayed with 20mL normal saline intraperitoneally before the peritoneum was sutured. The surgeon placed an intraperitoneal catheter with the catheter tip above the vaginal end while placing percutaneous drainage tube. Patients in both groups were routinely given flurbiprofen axel 50mg intravenously for analgesia. Local infiltration anesthesia was performed with 20mL 1% lidocaine at the incision area. In the control group, 0.9% normal saline was injected intraperitoneally with 10mL/h, and the total volume in the pump was 720mL. At the same time, patients in both groups were connected with intravenous controlled analgesia pump (PCIA) : sufentanil 100µg to 100mL normal saline, background dose of 2mL/h, single push injection of 0.5mL, locked for 15 minutes.
  Interventions: Procedure: intraperitoneal lidocaine analgesic or normal saline as control

INTERVENTIONS:
Procedure: intraperitoneal lidocaine analgesic or normal saline as control — Before the end of surgery, patients in the experimental group (L group) were extensively sprayed with 20mL (100mg) 0.5% lidocaine intraperitoneally before the peritoneum was sutured. The surgeon placed intraperitoneal catheter with the catheter tip above the vaginal end while placing percutaneous drainage tube. The intraperitoneal catheter was connected to the electronic analgesia pump, and the infusion of 0.5% lidocaine 10mL/h was interrupted from 1 to 72h after surgery, with a total volume of 720mL in the pump.

SUMMARY:
The main objective of this trial is to improve the postoperative analgesia effect and prognosis of patients with ovarian cancer after laparotomy surgery. This is a randomized, double-blind, controlled trial to evaluate analgesia and patient outcomes after local peritoneal anesthesia after surgery.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled clinical study. Sixty patients were expected to participate in a centralized randomized study method divided into two groups of 30 patients per group: the intraperitoneal analgesic group and the normal saline control group. Standard routine anesthesia was performed in both groups using the same method, and intravenous analgesia pump was routinely used in clinical use after surgery. The intraperitoneal analgesic group was continuously pumped with local anesthetics into the abdominal cavity, while the control group was pumped with normal saline. Visual analogue pain score (VAS), amount of remedial analgesia and use of analgesia pump were recorded at 1, 2, 4, 8, 12, 24, 36, 48, 60 and 72 hours after operation. Record the time when the patient began drinking and eating, and the time when gastrointestinal function (defecation or exhaust) recovered. The time of starting to walk on the ground (including the time of needing attendant assistance or not) and the time of meeting the standard of postoperative discharge preparation. Perioperative peripheral blood samples were collected for five times (T0 before anesthesia induction, T1 after tracheal extubation, T2 on the morning of the first postoperative day, T3 on the morning of the second postoperative day, and T4 on the morning of the third postoperative day), and inflammatory factors and tumor-related indicators were monitored. Adverse reactions were recorded. The prognosis of the patients was followed up 5 years after operation.

ELIGIBILITY:
Inclusion Criteria:

* The American Society of Anesthesiologists (ASA) rated them as grade I to II, aged 18 to 75 years.
* Patients undergoing elective laparotomy for ovarian cancer reduction (surgical resection includes the whole uterus with or without double adnexa, lymph node biopsy, dissection, appendectomy, etc.).

Exclusion Criteria:

* Suffering from mental illness or unable to cooperate with pain and related index scoring, unable to use automatic pump.
* Peritoneal infection existed before surgery
* Past history of arrhythmia
* Severe liver and kidney dysfunction existed before surgery
* Known allergy to local anesthetics
* Do not agree to participate in the research

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-18 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative analgesic use | Postoperative 72 hours
  Postoperative intravenous analgesia pump pressing time (recording the time by the electronic analgesia pump) and times (including effective and ineffective pressing times, recording by numbers), intravenous analgesia pump drug usage[sufentanil (µg)].

SECONDARY OUTCOMES:
Survival time (months) | Postoperative 5 years
  Postoperative survival time (months).
Disease free survival time (months) | Postoperative 5 years
  Time between surgery to cancer relapse (months).
Recurrence (yes/no, if yes ,record recurrence date) | Postoperative 5 years
  Whether the cancer relapse.
Postoperitive chronic pain duration (months) | Postoperative 5 years
  Postoperitive chronic pain duration (months), if present, record the location of the pain.

OTHER OUTCOMES:
Start drinking and eating time (hours) | During the time in the hospital. Up to 30 days post operation.
  Time when the patients start drinking and eating.
Time for recovery of gastrointestinal function (defecation or exhaust)(hours) | During the time in the hospital. Up to 30 days post operation.
  Time to the patients bowel movement recover.
The time for starting to walk. | During the time in the hospital. Up to 30 days post operation.
  Record the time of walk with attendant assistance (hours), and by theirselves____ (hours).
The standard time of postoperative discharge preparation ____ (hours) | During the time in the hospital. Up to 30 days post operation.
  Postoperative discharge preparation standards include: Walk independently, gastrointestinal function (to eat, drink, defecate) returned to normal, with oral analgesics, appropriate control without a mild pain, symptoms of nausea and vomiting, a local infection (redness, tenderness) or systemic infection, fever, c-reactive protein or increase white blood cell count), no other complications (bleeding, respiratory dysfunction, Deep vein thrombosis, etc.
Drainage tube and fluid. | During the time in the hospital. Up to 30 days post operation.
  Drainage tube removal time ____(hours), drainage volume ____(ml), drainage flow character ____(color/transparent/other).
Local anesthetic toxicity | During the time in the hospital. Up to 30 days post operation.
  Frequency of occurrence: Times of occurrence (number) The time of occurrence from surgery (hours) Symptoms (record) Treatment (record)
Nausea and vomiting: | During the time in the hospital. Up to 30 days post operation.
  Nausea and vomiting: Times of vomiting(number) The time of occurrence from surgery (hours) Treatment (record) Postoperative nausea score was recorded by numbers 0-3:0 = no nausea, 1= mild nausea and vomiting, which did not require drug treatment, 2= moderate nausea, which could be controlled by ondansetron, 3= severe nausea, which did not respond to ondansetron.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China